CLINICAL TRIAL: NCT01487200
Title: A Double-Blind, Randomized, Parallel Group, Active Comparator Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamic Effects (HPA Axis) of FX006 in Patients With Osteoarthritis of the Knee
Brief Title: Pharmacokinetic and Pharmacodynamic Study of FX006 in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FX006-2011-002
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Results first posted 2019-12-06 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis; knee; corticosteroid; intra-articular; injection
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — FX006; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- FX006 10mg (Experimental): Single 3 mL intra-articular (IA) injection Extended-release formulation
  Interventions: Drug: FX006 10 mg
- FX006 40mg (Experimental): Single 3 mL intra-articular (IA) injection Extended-release formulation
  Interventions: Drug: FX006 40 mg
- FX006 60 mg (Experimental): Single 3 mL intra-articular (IA) injection Extended-release formulation
  Interventions: Drug: FX006 60 mg
- TCA IR (40 mg) (Active Comparator): Single 1 mL intra-articular (IA) injection Immediate-release formulation
  Interventions: Drug: TCA IR 40

INTERVENTIONS:
Drug: FX006 10 mg — single 3 mL IA injection
  Arms: FX006 10mg
Drug: FX006 40 mg — single 3 mL IA injection
  Arms: FX006 40mg
Drug: FX006 60 mg — single 3 mL IA injection
  Arms: FX006 60 mg
Drug: TCA IR 40 — single 1 mL IA injection
  Other Names: Kenalog®-40; Kenacort-A 40; Triamcinolone Acetonide Crystalline Suspension (TAcs)
  Arms: TCA IR (40 mg)

SUMMARY:
The purpose of this study was to evaluate the safety, pharmacokinetics and pharmacodynamics of FX006 in patients with osteoarthritis of the knee.

DETAILED DESCRIPTION:
This study was a double-blind, randomized, parallel-group, active comparator design. The study was conducted in male and female patients ≥35 years of age with symptomatic OA of the knee.

Twenty-four (24) patients with knee OA were randomized (1:1:1:1) and treated with a single IA injection of either 10, 40, or 60 mg of FX006 or 40 mg of TCA IR.

Each patient was evaluated for a total of 6 weeks following a single IA injection. Following screening, safety, PK and pharmacodynamics (PD) were evaluated during one (1) 48-hour in-patient period (Day -1 to Day 2), two (2) 24-hour in-patient periods (Day 14-15 and Day 42-43) and seven (7) out-patient visits (Days 3, 4, 5, 8, 22, 29 and 36).

ELIGIBILITY:
Main Inclusion Criteria:

* Willingness and ability to comply with the study procedures and visit schedules and ability to follow verbal and written instructions
* Male or female >=35 years of age
* Diagnosis of unilateral or bilateral OA of the knee for at least 6 months prior to Screening with confirmation of OA according to American College of Rheumatology Criteria for Classification of Idiopathic OA of the Knee (clinical and radiological) based on an X-ray performed within 6 months prior to Screening or during the Screening period
* Body mass index (BMI) ≤ 40 kg/m2
* Willingness to abstain from use of the protocol-specified restricted medications

Main Exclusion Criteria:

* History of Reiter's syndrome, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, arthritis associated with inflammatory bowel disease, sarcoidosis or amyloidosis
* History of arthritides due to crystals (e.g., gout, pseudogout)
* History of infection in the index joint
* Clinical signs and symptoms of active knee infection or crystal disease of the index knee
* Presence of surgical hardware or other foreign body in the index knee
* Unstable joint (such as a torn anterior cruciate ligament)
* IA corticosteroid (investigational or marketed) in any joint within 3 months of Screening
* IA hyaluronic acid (investigational or marketed) in the index knee within 6 months of Screening
* Oral, inhaled or intranasal corticosteroids (investigational or marketed) within 1 month of Screening
* Prior arthroscopic or open surgery of the index knee within 12 months of Screening
* Planned/anticipated surgery of the index knee during the study period
* History of or active malignancy, with the exception of resected basal cell carcinoma, squamous cell carcinoma of the skin, or resected cervical atypia or carcinoma in situ within 5 years
* Insulin-dependent diabetes
* History of or active Cushing's syndrome
* Any other clinically significant acute or chronic medical conditions (e.g., uncontrolled diabetes)
* Skin breakdown at the knee where the injection would take place
* Women of child-bearing potential not using effective contraception or who are pregnant or nursing

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Bodick, MD, Study Director — Flexion Therapeutics
Locations (2):
- Australia (2):
  - Adelaide, South Australia
  - Perth, Western Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study took place at 2 centers, both located in Australia. Enrollment for this study took approximately 1.5 months.
Pre-assignment Details: Subjects were screened for eligibility within 14 days of being randomized
Groups:
- FX006 10mg: 5 subjects received FX006 10 mg as a single 3 mL IA injection.
- FX006 40mg: 7 subjects received FX006 40 mg as a single 3 mL IA injection.
- FX006 60 mg: 7 subjects received FX006 60 mg as a single 3 mL IA injection.
- TCA IR 40 mg: 5 subjects received commercially available triamcinolone acetonide (40 mg) as a single 1 mL IA injection.
Period: Overall Study
Arm/Group | FX006 10mg | FX006 40mg | FX006 60 mg | TCA IR 40 mg
Started | 5 | 7 | 7 | 5
Completed | 5 | 6 | 7 | 5
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- FX006 10mg; FX006 40mg; FX006 60 mg: Single 3 mL IA injection
- TCA IR (40 mg): Single 1 mL IA injection
- Total: Total of all reporting groups
Arm/Group | FX006 10mg | FX006 40mg | FX006 60 mg | TCA IR (40 mg) | Total
Number analyzed (Participants) | 5 | 7 | 7 | 5 | 24
Age, Continuous [Mean (Full Range); unit: years] | 63.2 [36 to 81] | 59.3 [49 to 75] | 64.9 [56 to 79] | 63 [53 to 76] | 62.5 [36 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 3 | 3 | 16
  Male | 1 | 1 | 4 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24-hour Weighted Mean Serum Cortisol
Description: The primary pharmacodynamic endpoint was change from baseline (pre-dose) to Day 1-2, Day 14-15 (Week 2) and Day 42-43 (Week 6) in 24-hour weighted mean serum cortisol. This is defined as AUC over the 0-24 hour measurement period divided by 24
Time Frame: Days 1-2, Days 14-15 (Week 2) and Days 42-43 (Week 6)
Measure: Least Squares Mean (95% Confidence Interval); unit: weighted mean serum cortisol (nmol/L)
Groups:
- TCA IR 40 mg: Single 1 mL IA injection
Arm/Group | FX006 10mg | FX006 40mg | FX006 60 mg | TCA IR 40 mg
Number analyzed (Participants) | 5 | 7 | 7 | 5
weighted mean serum cortisol (nmol/L)
  Change from BL to Days 1 to 2 | -7.7 [-38.4 to 38.3] | -42.7 [-59.2 to -19.4] | -62.2 [-73.2 to -46.8] | -59.0 [-72.6 to -38.6]
  Change from BL to Days 14 to 15 | -11.1 [-37.0 to 25.5] | -33.4 [-50.2 to -10.9] | -49.5 [-62.3 to -32.4] | -19.7 [-43.0 to 13.3]
  Change in BL to Days 42 to 43 | -9.0 [-26.2 to 12.3] | -18.0 [-32.2 to -0.7] | -11.8 [-26.1 to 5.4] | -4.8 [-22.7 to 17.4]

2. Primary Outcome: Characterize the Pharmacokinetic Profile of FX006 and TCA IR
Description: Concentrations below the limit of quantification of 50 pg/mL were treated as 0.
Time Frame: Day 1 (1, 2, 4, 6, 8, 12 and 24 hours post dose) and Days 3, 4, 5, 8, 15, 22, 29, 36 and 43
Population: PK population was to include all patients who received study drug and had at least one measurable concentration
Measure: Geometric Mean (Standard Deviation); unit: pg/mL
Arm/Group | FX006 10mg | FX006 40mg | FX006 60 mg | TCA IR 40 mg
Number analyzed (Participants) | 5 | 7 | 7 | 5
pg/mL
  1 hour postdose | 140.941 (0.4767) | 638.447 (0.6312) | 862.574 (0.6823) | 12268.835 (1.4681)
  2 hours postdose | 226.058 (0.2204) | 779.819 (0.6778) | 1164.013 (0.6772) | 14243.604 (1.5643)
  4 hours postdose | 280.406 (0.3637) | 860.476 (0.7088) | 1251.776 (0.7030) | 16282.659 (1.7765)
  6 hours postdose | 261.231 (0.4108) | 814.647 (0.7131) | 1182.925 (0.6952) | 14560.886 (1.7754)
  8 hours postdose | 249.298 (0.4640) | 748.962 (0.7898) | 1227.658 (0.6245) | 13543.427 (1.7347)
  12 hours postdose | 230.506 (0.5331) | 691.962 (0.7456) | 1127.476 (0.7841) | 10112.863 (1.6684)
  Day 2 (24 hrs post dose) | 242.764 (0.4037) | 763.568 (0.7423) | 1309.260 (0.5869) | 5421.894 (1.5196)
  Day 3 (48 hrs post dose) | 233.138 (0.3999) | 743.344 (0.7583) | 1294.042 (0.7645) | 2371.778 (1.1844)
  Day 4 (72 hrs post dose) | 224.987 (0.4904) | 675.086 (0.6930) | 1270.953 (0.7088) | 1310.061 (0.8301)
  Day 5 (96 hrs post dose) | 242.533 (0.3787) | 690.857 (0.7292) | 1252.021 (0.7097) | 822.243 (0.6002)
  Day 8 (168 hrs post dose) | 185.257 (0.5638) | 586.977 (0.7574) | 1070.823 (0.6322) | 235.938 (1.0814)
  Day 15 (336 hrs post dose) | 113.002 (0.5244) | 365.970 (0.7325) | 718.787 (0.5587) | 0.000 (0.000)
  Day 22 (504 hrs post dose) | 0.000 (0.000) | 238.529 (0.7026) | 521.843 (0.4563) | 0.000 (0.000)
  Day 29 (672 hrs post dose) | 0.000 (0.000) | 189.422 (0.6089) | 369.683 (0.4589) | 0.000 (0.000)
  Day 36 (840 hrs post dose) | 0.000 (0.000) | 0.000 (0.000) | 246.176 (0.3844) | 0.000 (0.000)
  Day 43 (1008 hrs post dose) | 0.000 (0.000) | 138.660 (0.6253) | 187.435 (0.3924) | 0.000 (0.000)

3. Secondary Outcome: Change From Baseline in 24-hour Urinary Free Cortisol Excretion
Time Frame: Baseline to Days 1-2, Baseline to Days 14-15 (Week 2) and Baseline to Days 42-43 (Week 6)
Population: Full Analysis Set (FAS) includes all observations from all patients who received a dose of study drug and provided a baseline observation and at least one post baseline observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: nmol/24h
Arm/Group | FX006 10mg | FX006 40mg | FX006 60 mg | TCA IR 40 mg
Number analyzed (Participants) | 5 | 7 | 7 | 5
nmol/24h
  Day 1 to 2 | 47.9 [-11.1 to 146.2] | -43.8 [-63.5 to -13.6] | -50.1 [-67.7 to -23.0] | -58.5 [-75.2 to -30.5]
  Day 14 to 15 | 13.0 [-25.3 to 70.8] | -42.4 [-59.3 to -18.3] | -59.0 [-72.0 to -40.0] | -14.7 [-43.9 to 29.6]
  Day 42 to 43 | 7.7 [-25.8 to 56.3] | -38.3 [-56.1 to -13.3] | -13.1 [-36.7 to 19.3] | -21.3 [-46.0 to 14.8]

4. Secondary Outcome: Total 24-hour Urinary Free Cortisol Excretion
Time Frame: Days 1-2, Days 14-15 (Week 2) and Days 42-43 (Week 6)
Population: FAS includes all observations from all patients who received a dose of study drug and provided a baseline observation and at least one post baseline observation.
Measure: Geometric Mean (Standard Deviation); unit: nmol/24h
Arm/Group | FX006 10mg | FX006 40mg | FX006 60 mg | TCA IR 40 mg
Number analyzed (Participants) | 5 | 7 | 7 | 5
nmol/24h
  Day 1 to 2 | 75.66 (1.112) | 29.94 (0.770) | 29.36 (0.490) | 18.77 (0.289)
  Day 14 to 15 | 57.14 (0.842) | 30.91 (0.590) | 26.46 (0.925) | 36.22 (0.962)
  Day 42 to 43 | 55.74 (0.715) | 34.62 (0.557) | 51.16 (0.499) | 36.38 (0.626)

5. Secondary Outcome: Change From Baseline to Each Measured Time Point Post-dose in Morning Serum Cortisol
Description: Least square mean difference against TCA IR 40 mg
Time Frame: Baseline to Days 2, 3, 4, 5, 8, 14, 15, 22, 29, 36, 42 and 43
Population: The full analysis set will include all observations from all patients who received any dose of FX006 and provide a baseline observation and at least one post baseline observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: nmol/L
Groups:
- TCA IR 40 mg: Single 1 mL IA injection of commercially available triamcinolone acetonide
Arm/Group | FX006 10mg | FX006 40mg | FX006 60 mg | TCA IR 40 mg
Number analyzed (Participants) | 5 | 7 | 7 | 5
nmol/L
  Day 2 | -30.2 [-68.9 to 57.1] | -42.3 [-71.1 to 15.1] | -78.2 [-89.1 to -56.4] | -85.4 [-93.5 to -67.1]
  Day 3 | -24.9 [-61.7 to 47.5] | -40.8 [-66.7 to 5.2] | -80.2 [-88.9 to -64.8] | -86.2 [-93.0 to -72.9]
  Day 4 | -13.9 [-58.1 to 77.3] | -37.1 [-66.0 to 16.4] | -77.2 [-87.7 to -57.8] | -73.1 [-86.9 to -44.6]
  Day 5 | -12.4 [-50.7 to 55.6] | -35.1 [-60.3 to 5.9] | -73.0 [-83.5 to -55.9] | -49.8 [-71.7 to -10.7]
  Day 8 | -29.8 [-50.1 to -1.1] | -37.4 [-53.2 to -16.1] | -61.7 [-72.2 to -47.4] | -8.6 [-35.1 to 28.8]
  Day 14 | -7.6 [-37.7 to 37.1] | -35.5 [-53.4 to -10.7] | -40.4 [-55.8 to -19.6] | -27.3 [-48.9 to 3.4]
  Day 15 | -24.4 [-48.2 to 10.4] | -28.1 [-47.9 to -0.7] | -46.4 [-61.2 to -26.0] | -8.3 [-37.2 to 34.0]
  Day 22 | 3.3 [-26.6 to 45.2] | -28.5 [-46.5 to -4.4] | -14.4 [-36.0 to 14.6] | -11.3 [-36.9 to 24.9]
  Day 29 | -4.5 [-26.8 to 24.5] | -21.1 [-37.1 to -1.1] | -6.3 [-25.3 to 17.5] | 0.8 [-22.7 to 31.5]
  Day 36 | -6.4 [-33.5 to 31.7] | -19.5 [-39.8 to 7.7] | -3.0 [-27.6 to 29.8] | 11.7 [-20.7 to 57.2]
  Day 42 | -18.3 [-47.8 to 27.7] | -27.0 [-49.5 to 5.4] | -19.1 [-42.4 to 13.6] | -21.4 [-47.3 to 17.1]
  Day 43 | -22.1 [-39.1 to -0.3] | -14.9 [-32.2 to 6.8] | -13.4 [-29.8 to 6.9] | 3.0 [-19.5 to 31.9]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from post injection on Day 1 through Day 43.
Arm/Group | FX006 10mg | FX006 40mg | FX006 60 mg | TCA IR 40 mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/7 | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7 | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 4/5 | 7/7 | 6/7 | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FX006 10mg (N=5) | FX006 40mg (N=7) | FX006 60 mg (N=7) | TCA IR 40 mg (N=5)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site haematoma (General disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 3 (3) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other